CLINICAL TRIAL: NCT03098758
Title: Pilot Study of Comparative Molecular Analysis CK20, CEA and BER-EP4 in Peritoneal Washing Citology for Locally Advanced Gastric Cancer and Their Ability to Predict Peritoneal Dissemination
Brief Title: Molecular Analysis in Peritoneal Washing Citology for Locally Advanced Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Alexis Luna, MD PhD, Corporacion Parc Tauli
Other Study IDs: CIRPT_AL2017_1
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Gastric Cancer; Polymerase Chain Reaction
Keywords: Polymerase Chain Reaction; gastric cancer; citology; peritoneal washing; CK20; CEA; BER-EP4
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — gastric cancer cells in peritoneal washing
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gastric carcinoma is a disease with a high mortality. Peritoneal washing cytology has a recognized prognostic utility. However sensibility of this study is not appropriate. Studies with PCR (polymerase chain retrotranscription) can increase sensibility and accurate staging information.

Objective: To analyze the sensibility and specificity of the expression of CK20, CEA and Ber-EP4 with PCR technique in peritoneal washings of advanced gastric carcinoma without clinical evidence of peritoneal carcinomatosis.

Methodology: Retrotranscription analysis (RT-PCR) and quantitative PCR (qPCR) of CK20, CEA and Ber-EP4 in peritoneal washing. Test the feasibility of qPCR with this new marker (Ber-EP4). Comparison of the results with data obtained with conventional cytology. Study of peritoneal recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients with resectable advanced gastric cancer
* Informed consent

Exclusion Criteria:

* Macroscopic peritoneal carcinomatosis
* Non operable patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced gastric cancer without macroscopic peritoneal carcinomatosis
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-05-08 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
specific markers in peritoneal cells | during surgical intervention
  Detection of CK20, CEA and BER-EP4 by PCR technique in peritoneal washing of advanced gastric cancer

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Luna, MD PhD, Principal Investigator — Corporación Parc Taulí
Locations (1):
- Parc Tauli Hospital Universitari, Sabadell, Barcelona, Spain